CLINICAL TRIAL: NCT05300126
Title: HypnoPal : a Mixed Method Study of a Home Based Hypnosis Intervention for Palliative Care Patients and Their Relatives
Brief Title: Brief Hypnosis Intervention for Palliative Care Patients and Their Relatives.
Acronym: HypnoPal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Teike Luthi Fabienne, Principal investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-02193
Record Dates: First submitted 2022-01-26; First posted 2022-03-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Palliative Care; Hypnosis; Home
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual care (Experimental): No hypnosis session are proposed
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — Four sessions of 15 minute hypnosis, based on standardised script, focused on symptom management for the patients and of resource development for relatives.

SUMMARY:
The study objective is to assess the feasibility of hypnosis sessions for palliative care patients in home care and of their relatives. The intervention consists of four 15-minute hypnosis sessions for the patients and for one family member, taking place at the patient's home. Recordings will be given to practice self-hypnosis.

DETAILED DESCRIPTION:
The primary outcome of this study is to assess the feasibility of a home based hypnosis intervention, targeting the management of symptoms (e.g. pain, anxiety) of palliative care patients and the reinforcement of a positive skill for their relatives (e.g. acceptance, relaxation), as well as the development of their respective self-hypnosis practice.

The two secondary outcomes are: i) to understand what the needs of palliative care patients and their relatives are in relation to complementary medicine and ii) to understand the process of integration of complementary medicine into usual care by looking at how this takes place for the participants to the intervention as well as for other palliative care patients who resort to using complementary medicine (not limited to hypnosis).

This is a mixed-methods study combining quantitative and qualitative data in a convergent design. The convergent design, derived from the pragmatic paradigm, involves the independent collection and analysis of quantitative and qualitative data. The results are then merged in order to compare and/or combine them and thus provide a broader understanding of the issue being studied.

For the intervention, participants will be recruited by a community mobile palliative care team. They will be screened by the study team to ensure they fulfil the inclusion criteria. If eligible and after informed consent is obtained, an assessment of the cognitive function will be performed. The patients will then recruit one of their relatives for participation to the study.

For the secondary outcomes, participants will be healthcare professionals working in palliative care setting and using complementary medicine in their daily practice and also patients using complementary medicine but who do not participate at the interventional part of this study.

ELIGIBILITY:
Inclusion Criteria :

* adults ≥18 years
* followed by a mobile palliative care team
* expressed symptom such as: pain, dyspnea, sleep disturbance or anxiety at a score of ≥ 3/10 at inclusion
* interest in managing symptoms with hypnosis

Exclusion Criteria :

* inability to communicate in French without a translator
* severe cognitive impairment
* severe hearing impairment
* acute psychiatric or somatic decompensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Expectations of hypnosis in terms of personal benefits assessed by VAS | Change from baseline hypnosis expectations at 4 weeks
  Measured at Baseline - Question: how well do you expect this treatment to work for you (VAS: 0: no effect at all to 10: full relief)
Acceptance rate of the intervention assessed by descriptive numeric data | 1 year
  How many times the intervention was proposed and how many patients and relatives were interested in and had participated
Number of sessions carried out and their duration assessed by descriptive numeric data | 1 year
  For each patient and relatives the number of sessions and duration of each session is collected
Symptom intensity assessed by Edmonton Symptom Assessment System | Change from symptom intensity at 4 weeks
  Nine symptoms are assessed by VAS: 0: no symptom at all to 10: maximal intensity
Quality of life assessed by VAS | Change from baseline quality of life at 4 weeks
  The global quality of life is assessed by VAS 0: minimal to 10: maximal
Comfort assessed by VAS | Change from baseline comfort at 4 weeks
  The global comfort is assessed by VAS 0: minimal to 10: maximal
The main symptom intensity assessed by VAS | 15 minutes
  The main symptom present before the hypnosis session is assessed by VAS: 0: no symptom at all to 10: maximal intensity
Satisfaction and needs assessed by semi structured interview | 4 weeks
  To globally understand the experience of the hypnosis intervention

SECONDARY OUTCOMES:
Needs and integration assessed by semi structured interview | through study completion, an average of 1 year
  To assess the needs of this specific population regarding the integrative medicine and the integration of complementary medicine into routine care by interviewing professionals, patients and relatives

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Teike Lüthi, PhD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Teike Lüthi Fabienne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No